CLINICAL TRIAL: NCT03940495
Title: A Prospective Study to Evaluate Whether Serum Kisspeptin is a Marker Predictive of the First Trimester Miscarriage of Women Who Conceive in IVF
Brief Title: Serum Kisspeptin: a Predictive Marker of Miscarriage or Not?
Status: Completed | Type: Observational
Sponsor: ShangHai Ji Ai Genetics & IVF Institute (Other)
Responsible Party: Sponsor
Other Study IDs: JIAI 2019-04
Record Dates: First submitted 2019-05-04; First posted 2019-05-07 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2020-04

CONDITIONS: Miscarriage
MeSH Terms: conditions — Abortion, Spontaneous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood serum for hCG level is performed 14 days after embryo transfer i.e. week 4. If the serum hCG level is >10IU/L, the women are considered pregnant and serum will be saved and checked for kisspeptin level, Blood test is repeated at 5 weeks and 6 weeks
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective observational study. Eligible women undergo ART treatment in our centre will be recruited for the study and each woman will only be included in the study once. Informed written consent will be obtained. Blood serum for hCG level is performed 14 days after the embryo transfer i.e. week 4. If the serum hCG level is >10IU/L, the women are considered pregnant and blood will be saved and checked for kisspeptin level, Another blood test is repeated 1 week later i.e. week 5. A transvaginal ultrasound and blood test will be performed 1 week later i.e. week 6 to confirm the fetal viability and the number of gestational sacs and locate the pregnancy.

Blood for hCG and kisspeptin levels are checked at weeks, 4, 5 and 6. Ultrasound will be performed at gestational 8 weeks and 11 weeks. They will be referred for antenatal care when the pregnancy is confirmed on-going at 11 weeks.

The purpose is to determine whether serum kisspeptin level in women who conceive in IVF is associated with an increased risk in first trimester miscarriage and compare with serum hCG level in the prediction of the first trimester miscarriage.

ELIGIBILITY:
Inclusion Criteria:

* Women who have a positive pregnancy test following IVF or frozen-thawed transfer

Exclusion Criteria:

* Women with renal failure are excluded due to assay interference with kisspeptin measurement

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Eligible women undergo ART treatment in our centre Shanghai JiAi Genetics & IVF Institute will be recruited for the study and each woman will only be included in the study once. Informed written consent will be obtained.
Sampling Method: Probability Sample
Enrollment: 182 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Early miscarriage loss | 10 weeks
  defined as intrauterine pregnancy loss at less than 10 weeks' gestation as identified by ultrasound, including identification of empty sac, miscarriage, yolk sac miscarriage and embryonic miscarriage

SECONDARY OUTCOMES:
Biochemical pregnancy | 8 weeks
  defined as pregnancy demise based on decreasing serum or urinary beta-HCG levels, without ultrasound visualization
Positive hCG level | 4 weeks
  conception is defined with the result of serum β-hCG ≥10 mIU/mL.

CONTACTS AND LOCATIONS:
Overall Officials: XIAOXI SUN, PHD, Study Director — Shanghai JiAi Genetics & IVF Institute, China
Locations (1):
- ShangHai JIAI Genetics&IVF Institute, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results after deidentification (text, tables, figures, and appendices) and study protocol will be shared. Data will be available when beginning 3 months and ending 5 years following article publication. To achieve aims in the approved proposal, researchers who provide a methodologically sound proposal will be shared with.Data will be made available by the following way. Proposals should be directed to lihe198900@163.com. And data are available for 5 years at a third party website (link to be included after the article publication).

REFERENCES:
- [Background] Kolte AM, Bernardi LA, Christiansen OB, Quenby S, Farquharson RG, Goddijn M, Stephenson MD; ESHRE Special Interest Group, Early Pregnancy. Terminology for pregnancy loss prior to viability: a consensus statement from the ESHRE early pregnancy special interest group. Hum Reprod. 2015 Mar;30(3):495-8. doi: 10.1093/humrep/deu299. Epub 2014 Nov 5. PMID 25376455
- [Background] Ammon Avalos L, Galindo C, Li DK. A systematic review to calculate background miscarriage rates using life table analysis. Birth Defects Res A Clin Mol Teratol. 2012 Jun;94(6):417-23. doi: 10.1002/bdra.23014. Epub 2012 Apr 18. PMID 22511535
- [Background] Horne AW, McBride R, Denison FC. Normally rising hCG does not predict live birth in women presenting with pain and bleeding in early pregnancy. Eur J Obstet Gynecol Reprod Biol. 2011 May;156(1):120-1. doi: 10.1016/j.ejogrb.2011.01.013. Epub 2011 Feb 18. No abstract available. PMID 21334129
- [Background] Jayasena CN, Abbara A, Izzi-Engbeaya C, Comninos AN, Harvey RA, Gonzalez Maffe J, Sarang Z, Ganiyu-Dada Z, Padilha AI, Dhanjal M, Williamson C, Regan L, Ghatei MA, Bloom SR, Dhillo WS. Reduced levels of plasma kisspeptin during the antenatal booking visit are associated with increased risk of miscarriage. J Clin Endocrinol Metab. 2014 Dec;99(12):E2652-60. doi: 10.1210/jc.2014-1953. PMID 25127195
- [Background] Sullivan-Pyke C, Haisenleder DJ, Senapati S, Nicolais O, Eisenberg E, Sammel MD, Barnhart KT. Kisspeptin as a new serum biomarker to discriminate miscarriage from viable intrauterine pregnancy. Fertil Steril. 2018 Jan;109(1):137-141.e2. doi: 10.1016/j.fertnstert.2017.09.029. PMID 29307393
- [Derived] Li H, Zhang W, Sun X. A prospective study to evaluate whether serum kisspeptin is a marker predictive of the first-trimester miscarriage of women who conceive in IVF. J Assist Reprod Genet. 2024 Jan;41(1):79-85. doi: 10.1007/s10815-023-02974-x. Epub 2023 Nov 8. PMID 37935913